CLINICAL TRIAL: NCT05224219
Title: Modified Preloaded System for Renal Arteries in Fenestrated Endografting
Brief Title: Modified Preloaded System for Renal Arteries in Fenestrated Endografting (MPSRA)
Acronym: MPSRA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Enrico Gallitto, Principal Investigator, University of Bologna
Other Study IDs: MPSRA
Record Dates: First submitted 2022-01-04; First posted 2022-02-04 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Juxtarenal Aortic Aneurysm; Thoracoabdominal Aortic Aneurysm; Pararenal Aortic Aneurysm; Aortic Aneurysm, Thoracoabdominal; Dissection Aortic Aneurysm; Penetrating Aortic Ulcer; Endoleak; Pseudoaneurysm
MeSH Terms: conditions — Aortic Aneurysm, Thoracoabdominal; Aortic Dissection; Penetrating Atherosclerotic Ulcer; Endoleak; Aneurysm, False

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Advanced Endovascular repair of aneurysms and dissections involving thoraco-abdominal (type I-IV) and complex abdominal (juxta and para-renal) aorta is a ground-gaining procedure allowing favorable results in high surgical risk patients. The availability of iliac vessels navigation and the major role of lower leg perfusion in order to decrease the risk of spinal cord ischemia during these complex procedures, led to the development of devices with lower sheaths sizes and to the improvement of the technique with preloaded devices for visceral vessels in order to navigate in hostile anatomies or when an iliac access is not available. The aim of the study is to evaluate in a prospective single center observational setting, the outcomes, safety and efficacy of the modified preloaded system for renal arteries in fenestrated endografting in the routine treatment of paravisceral and thoraco-abdominal aortic pathologies.

DETAILED DESCRIPTION:
Thoracoabdominal aortic aneurysm (TAAA) and complex abdominal aortic aneurysms (AAA) represents an evolving pathology that involves to varying degrees both the descending thoracic aorta and the abdominal aorta. These aneurysms, according to their localization and involvement in the thoracic and abdominal aorta, have been classified according to Crawford into 4 groups (I-IV) for the TAAA and in pararenal/juxtarenal (p/j-AAA) for AAA when a standard endovascular repair is not possible.

The prevalence of these pathologies is currently not well known, but high mortality rates are reported in the population carrying TAAAs and j/p-AAAs that have not undergone surgical treatment, most of which are due to aortic rupture.

Among of the main complications related to TAAA endovascular repair and to complex AAA we can account spinal cord ischemia, lower leg ischemia and logo-operative times, that all can contribute to decrease overall technical and clinical success.

A particular subgroup of TAAAs is represented by post-dissection thoracoabdominal aneurysms (PDTAA), which represents an evolving pathology and one of the main chronic complications in outcomes of acute chronic dissection. In these particular subset of patients, as well as in patient with highly calcified and hostile accesses, the risk of post-operative spinal cord ischemia is higher and the availability of both iliac access navigability is not always possible, leading to technical failure, intraoperative complications and need for adjunctive invasive procedures in high surgical risk patients.

The fenestrated and branched endoprostheses (F/B-EVAR) represent a technology that is now firmly used for the treatment of thoraco-abdominal degenerative aneurysmal pathology in superspecialized centers. Recently, the technology with F/B-EVAR has also been used in the treatment of PDTAA, IMH and PAU, showing satisfactory results. This experience has been carried out in some centers, in the absence, however, of a wider and generalized experience. All these type of endografts are custom-made devices, requiring therefore a lading time for production and delivering before being implanted into the specific patient.

In order to overcome main drawbacks of these procedures, such us long operating time due to fenestrations and vessels cannulation, to avoid bilateral lower limbs ischemia due to large bore introducer sheaths and to accomplish successful delivery even in patient without navigability of both iliac accesses, a modified preloaded system for renal arteries has been developed by Cook (Cook Medical, Bloomington, IN, USA).

The aim of the study is to evaluate in a prospective single center study observational setting, the outcomes, safety and efficacy of the modified preloaded system for renal arteries developed by Cook Medical with bi-port handle system in the field of fenestrated endografting during the routine treatment of thoraco-abdominal and paravisceral abdominal aortic pathologies.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of thoraco-abdominal or complex abdominal aortic aneurysm confirmed by a Computed tomography Angiography (CTA).
* Etiologies will be degenerative aneurysms, inflammatory aneurysms, chronic post-dissectional aneurysms, penetrating aortic ulcers, failure of prior surgical or endovascular repair.
* Elective aneurysmal repair of patient with maximum diameter greater than 55 mm, or fast growing, or symptomatic aneurysms.
* Endovascular repair performed using custom-made fenestrated and/or branched endografting with presence of modified preloaded system with modified handle and preloaded catheters for visceral vessels cannulation.

Exclusion Criteria:

* Patients submitted to advanced fenestrated and branched endovascular repair with other grafts besides the Cook Medical custom-made endograft or without modified handle preloaded delivery system.
* Physician-modified devices
* Patient treated with hybrid and/or open technique as well as parallel grafts (such as chimney/snorkel/periscope)
* Patient treated as emergent/urgent patients or aneurysmal rupture
* Patient who can not wait for the lead time required for endograft production and delivery.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All elective patients treated in a single center institution, with the standard of care for thoraco-abdominal and para-juxta-renal abdominal aortic aneurysms using fenestrated/branched custom-made endograft developed by Cook Medical with modified preloaded system for renal arteries.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Technical Success | Intra-operative final completion angiography.
  Successful deployment of custom-made modified endograft, target vessel patency and aneurysm exclusion, in absence of intra-operative mortality.
Mortality | Within the first 30-days from the procedure.
  Assessment of mortality related to procedure

SECONDARY OUTCOMES:
Cardiovascular Adverse Events | Within the first 30-days from the procedure.
  Cardiopulmonary and renal events related to the procedure.
Neurologic Adverse Events | Within the first 30-days from the procedure.
  Incidence of Spinal Cord Ischemia (transient/permanent) and Stroke
Vessel Instability | Within the first 30-days from the procedure.
  Target vessel patency and absence of stenosis, endoleak, occlusion, need for reintervention
Rate of early reintervention | Within the first 30-days from the procedure.
  Any re-intervention needed after the type of procedure and the specific reason
Overall Survival | Through study completion, an average of 1 year.
  Assessment of mortality in the post-operative period
Aorta Related Survival | Through study completion, an average of 1 year.
  Assessment of mortality in the post-operative period related to aortic procedure or aortic related death.
Freedom from reintervention | Through study completion, an average of 1 year.
  Time from procedure to the first aortic related/procedure related reintervention
Freedom from Vessel Instability | Through study completion, an average of 1 year.
  Target vessel patency and absence of stenosis, endoleak, occlusion, need for reintervention
Freedom from Major Endoleaks | Through study completion, an average of 1 year.
  Time from procedure to the presence of high-flow endoleak (TypeI/III) and from endoleak that required reintervention

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bologna, Bologna, Emilia-Romagna, Italy

REFERENCES:
- [Result] Gallitto E, Faggioli G, Spath P, Pini R, Mascoli C, Ancetti S, Stella A, Abualhin M, Gargiulo M. The risk of aneurysm rupture and target visceral vessel occlusion during the lead period of custom-made fenestrated/branched endograft. J Vasc Surg. 2020 Jul;72(1):16-24. doi: 10.1016/j.jvs.2019.08.273. Epub 2020 Feb 13. PMID 32063442
- [Result] Gallitto E, Gargiulo M, Faggioli G, Pini R, Mascoli C, Freyrie A, Ancetti S, Stella A. Impact of iliac artery anatomy on the outcome of fenestrated and branched endovascular aortic repair. J Vasc Surg. 2017 Dec;66(6):1659-1667. doi: 10.1016/j.jvs.2017.04.063. Epub 2017 Sep 6. PMID 28888759
- [Result] Maurel B, Resch T, Spear R, Roeder B, Bracale UM, Haulon S, Mastracci TM. Early experience with a modified preloaded system for fenestrated endovascular aortic repair. J Vasc Surg. 2017 Apr;65(4):972-980. doi: 10.1016/j.jvs.2016.09.045. PMID 28342523
- [Result] Spanos K, Kolbel T, Kubitz JC, Wipper S, Konstantinou N, Heidemann F, Rohlffs F, Debus SE, Tsilimparis N. Risk of spinal cord ischemia after fenestrated or branched endovascular repair of complex aortic aneurysms. J Vasc Surg. 2019 Feb;69(2):357-366. doi: 10.1016/j.jvs.2018.05.216. Epub 2018 Oct 29. PMID 30385148
- [Result] Bertoglio L, Loschi D, Grandi A, Melloni A, Bilman V, Melissano G, Chiesa R. Early Limb Reperfusion Using Routinely Preloaded Fenestrated Stent-graft Designs for Complex Endovascular Aortic Procedures. Cardiovasc Intervent Radiol. 2020 Dec;43(12):1868-1880. doi: 10.1007/s00270-020-02596-1. Epub 2020 Jul 19. PMID 32686037